CLINICAL TRIAL: NCT02018211
Title: Neuromuscular Electrical Stimulation Via the Peroneal Nerve Reduces Muscle Soreness Following Intermittent Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Collaborators: Loughborough University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FK-Sport-001; Loughborough (Other: Loughborough)
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: delayed onset muscle soreness; muscle damage; muscle function; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental group (Experimental): All participants performed a modified version of the Loughborough Intermittent Shuttle Test (LIST; Nicholas et al, 2000), an exercise protocol designed to simulate the activity pattern characteristics of intermittent sports such as soccer. The LIST was performed on three occasions, at the same time of day, each separated by approximately four weeks. Following each exercise trial, one of three recovery interventions were applied, the order of which were randomly allocated.
  Interventions: Other: control; Device: graduated compression socks; Device: neuromuscular electrical stimulation device

INTERVENTIONS:
Other: control — passive recovery following exercise test
Device: graduated compression socks — graduated compression socks worn after test exercise
Device: neuromuscular electrical stimulation device — neuromuscular electrical stimulation device worn after test exercise
  Other Names: firefly device

SUMMARY:
Numerous techniques are reported to enhance recovery following intense exercise, however there is equivocal support for such claims. A novel technique of neuromuscular electrical stimulation (NMES) via the peroneal nerve has been shown to augment limb blood flow which could enhance recovery following exercise. The present study examined the effects of NMES, compared to graduated compression socks on muscle soreness, strength, and markers of muscle damage and inflammation following intense intermittent exercise.

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* currently playing intermittent sports (such as soccer, field hockey, rugby)
* currently representing their respective sports at either university, county, national or international levels

Exclusion Criteria:

* unhealthy males
* not currently playing intermittent sports (such as soccer, field hockey, rugby)
* not currently representing their respective sports at either university, county, national or international levels
* individuals indicating a history of cardiovascular, metabolic or haematological disorders
* participants reporting a sedentary lifestyle of less than three 30-min physical activity sessions per week

Ages: 20 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Perceived muscle soreness (PMS) | 72hrs
  perceived muscle soreness (PMS), often referred to as delayed onset muscle soreness (DOMS)

SECONDARY OUTCOMES:
muscle strength | 72hrs

OTHER OUTCOMES:
measurement of CK and LDH activity and IL-6, CRP and TBAR concentrations | 72 hrs
  markers of muscle damage and inflammation following intense intermittent exercise

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sport, Exercise and Health Sciences, Loughborough, Leicestershire, United Kingdom

REFERENCES:
- [Result] Ferguson RA, Dodd MJ, Paley VR. Neuromuscular electrical stimulation via the peroneal nerve is superior to graduated compression socks in reducing perceived muscle soreness following intense intermittent endurance exercise. Eur J Appl Physiol. 2014 Oct;114(10):2223-32. doi: 10.1007/s00421-014-2943-5. Epub 2014 Jul 11. PMID 25011496